CLINICAL TRIAL: NCT00342862
Title: Assessment and Tracking of Long-Term Alefacept (LFA-3/IgG1 Fusion Protein) Pregnancy Exposure Registry
Brief Title: AMEVIVE® Pregnancy Registry
Status: Terminated | Type: Observational
Why Stopped: The Sponsor has made a decision, driven by business needs, to cease promotion, manufacturing, distribution and sales of Amevive
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 0485-CL-0002; C-739; NCT00168675 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Pregnancy
Keywords: Pregnancy; Amevive; alefacept; Registry; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Alefacept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1. Amevive Exposure: Pregnant women with psoriasis exposed to AMEVIVE® at any point within 8 weeks prior to conception, or at any time during pregnancy, where the outcome of the pregnancy is unknown prospectively
  Interventions: Drug: Amevive exposure

INTERVENTIONS:
Drug: Amevive exposure — Observational
  Other Names: alefacept; ASP0485

SUMMARY:
This is an observational, exposure-registration and follow-up study, to be conducted in the United States (US). The AMEVIVE® Pregnancy Exposure Registry is designed to monitor pregnant subjects and fetuses exposed to AMEVIVE® in order to detect any potential increase in the risk of major birth defects.

The AMEVIVE® Pregnancy Exposure Registry is sponsored by Astellas Pharma Global Development and will be managed by INC Research. The Registry will be monitored by an independent Advisory Committee of external experts in relevant specialties of teratology, epidemiology, maternal and fetal medicine, and infectious disease medicine (external member details available upon request).

DETAILED DESCRIPTION:
Prospective reports will be collected from pregnant subjects, health care provider (HCP), or Astellas Product Safety Management staff. Data from the pregnant subjects will be collected at 4 to 5 months of pregnancy by telephone interviews with the Registry. The Registry will also contact the subject at 2 months and 12 months after the estimated delivery date (EDD) for post-natal & pediatric follow-up. The Registry will confirm the information collected from the subject with the HCP by telephone interviews with the Registry, forms mailed/faxed to the Registry, electronic forms/queries sent to the Registry, or a combination of these methods. If a live birth is reported, the infant's HCP will be contacted for the Pediatric Follow-Up at 2 months and 12 months of age. If a birth defect is reported, targeted follow-up will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Have been exposed to AMEVIVE® within 8 weeks prior to conception or at any time during pregnancy
* Provide sufficient information to determine that the pregnancy is prospectively registered (i.e., the outcome of pregnancy must be unknown prospectively)
* Provide verbal consent to participate in the Registry, and
* Verbally provide the contact information for herself, her healthcare provider (HCP), and the infant's HCP (if applicable)

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women with psoriasis exposed to AMEVIVE® at any point within 8 weeks prior to conception, or at any time during pregnancy, where the outcome of the pregnancy is unknown prospectively
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2003-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Evaluate pattern or increase in major birth defects in children of women w/ psoriasis who were exposed to AMEVIVE® at any time within the 8 wks prior to conception, or at any time during pregnancy, where outcome of the pregnancy is unknown prospectively | At month 4 to 5 of pregnancy; At 2 months and 12 months post estimated delivery date

SECONDARY OUTCOMES:
To evaluate the number of live born infants versus fetal loss in pregnant women exposed to AMEVIVE® | At 2 months post estimated delivery date
To evaluate gestational age, body weight, gender, head circumference, and body length in live born infants exposed to AMEVIVE® | At 2 months post estimated delivery date
To evaluate appearance, pulse, grimace, activity, and respiration (APGAR) scores at 1 and 5 minutes of age in live born infants exposed to AMEVIVE® | At 2 months post estimated delivery date
To evaluate hospitalizations for infection in live born infants exposed to AMEVIVE® | At 2 months and 12 months post estimated delivery date
To evaluate clinically significant infections with unusual organisms, not requiring hospitalization in live born infants exposed to AMEVIVE® | At 2 months and 12 months post estimated delivery date
To evaluate malignancies in live born infants exposed to AMEVIVE® | At 2 months and 12 months post estimated delivery date

CONTACTS AND LOCATIONS:
Overall Officials: Vice President Medical Affairs, Study Director — Astellas Pharma Global Development
Locations (1):
- INC Research, Wilmington, North Carolina, United States